CLINICAL TRIAL: NCT04312100
Title: Sequential Oxygen Therapy Strategy for Patients With COVID-19
Acronym: SOTSPC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SOT-C
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus Disease-2019
Keywords: SARS-CoV-2; COVID-19; oxygen treatment
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Mild cases with conventional oxygen therapy: COVID-19 patients who were considered mild cases will receive conventional oxygen therapy in addition to standard treatment
  Interventions: Other: oxygen treatment
- Moderate/Severe cases with nasal high flow oxygen inhalation: COVID-19 patients who were considered Moderate/Severe cases will receive nasal high flow oxygen inhalation in addition to standard treatment
  Interventions: Other: oxygen treatment
- Moderate/Severe cases with non-invasive ventilation: COVID-19 patients who were considered Moderate/Severe cases will receive non-invasive positive pressure ventilation in addition to standard treatment
  Interventions: Other: oxygen treatment

INTERVENTIONS:
Other: oxygen treatment — different kinds of oxygen treatments will be given to patients according to their state of illness

SUMMARY:
All patients with COVID-19 were divided into three groups according to their illness: mild patient who receive conventional oxygen therapy, severe patients who receive nasal high flow oxygen inhalation or non-invasive positive pressure ventilation，all the oxygen therapy will be used as part of the standard of care. Each group will enroll 10 patients, the treatment of all patients will be continuously optimized during observation, and the incidence of respiratory failure, intubation rate, 28 day mortality rate, ICU hospitalization days, etc will be recorded and analyzed so to optimize the treatment time window of sequential oxygen therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COVID-19

  * Aged between 18-75 years;

    * Willing to sign the informed consent voluntarily.

Exclusion Criteria:

* Patients with active tuberculosis, idiopathic pulmonary fibrosis, bronchial asthma, bronchiectasis, pulmonary embolism, chronic respiratory failure or other serious respiratory diseases; ② patients with serious cardiovascular and cerebrovascular diseases (malignant arrhythmia, unstable angina, acute myocardial infarction, cardiac function grade 3 or above, stroke, cerebral hemorrhage, etc.); ③ Patients with serious hepatorenal diseases (serious liver diseases refer to cirrhosis, portal hypertension and varicose bleeding, and serious kidney diseases include dialysis and kidney transplantation); ④ tumor patients who have undergone resection, radiotherapy and chemotherapy within 5 years; ⑤ patients who have difficulty in activity due to neuromuscular diseases; ⑥ patients with serious arthritis; ⑦ patients with serious peripheral vascular diseases; ⑧ Pregnant and lactating women; ⑨ with severe cognitive and mental disorders; ⑩ the clinical researchers who were participating in other interventions within one month before selection;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients diagnosed with COVID-19 will be enrolled, diagnosis will depend on RT-PRC provided by China CDC
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of respiratory failure | 28 day
  Incidence of respiratory failure at day 28 after enrollment

SECONDARY OUTCOMES:
28 day mortality rate | 28 day
  mortality rate at day 28 after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoju Zhang, PhD, Principal Investigator — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan JF, Lau SK, To KK, Cheng VC, Woo PC, Yuen KY. Middle East respiratory syndrome coronavirus: another zoonotic betacoronavirus causing SARS-like disease. Clin Microbiol Rev. 2015 Apr;28(2):465-522. doi: 10.1128/CMR.00102-14. PMID 25810418
- [Background] Wu P, Hao X, Lau EHY, Wong JY, Leung KSM, Wu JT, Cowling BJ, Leung GM. Real-time tentative assessment of the epidemiological characteristics of novel coronavirus infections in Wuhan, China, as at 22 January 2020. Euro Surveill. 2020 Jan;25(3):2000044. doi: 10.2807/1560-7917.ES.2020.25.3.2000044. PMID 31992388
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4369385/